CLINICAL TRIAL: NCT05027230
Title: A Phase Ib/II,Multi-center, Open, Multiple-dose Design to Evaluate the Safety,Tolerability and Efficacy of STSP-0601 for Injection in Patients With Inhibitory Hemophilia
Brief Title: A Safety and Efficacy Study of STSP-0601 in Adult Patients With Hemophilia A or B With Inhibitor
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STSP-0601-02
Record Dates: First submitted 2021-08-25; First posted 2021-08-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consecutive doses of low-dose of STSP-0601 (Experimental)
  Interventions: Drug: STSP-0601 for Injection
- Consecutive doses of high-dose of STSP-0601 (Experimental)
  Interventions: Drug: STSP-0601 for Injection

INTERVENTIONS:
Drug: STSP-0601 for Injection — A multiple-dose design to evaluate the safety,tolerability and efficacy of two doses of STSP-0601 for injection in patients with inhibitory hemophilia
  Arms: Consecutive doses of low-dose of STSP-0601
Drug: STSP-0601 for Injection — A multiple-dose design to evaluate the safety,tolerability and efficacy of two doses of STSP-0601 for injection in patients with inhibitory hemophilia
  Arms: Consecutive doses of high-dose of STSP-0601

SUMMARY:
This study will assess the safety and efficacy of multiple-dose of STSP-0601 for the treatment of bleeding episodes in hemophilia A or B patients with inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤age≤65 years of age,male.
* Hemophilia A or B patients with inhibitors.
* Received hemostatic treatment with investigational drug, or to undergo minor surgical or other invasive procedures (Only for phase 2. Minor surgical procedures: procedures without general anesthesia and the wounds are easy to observe).
* Peak historical inhibitor titer ≥ 5 BU and a positive inhibitor test when enrolled.
* Establish proper venous access.
* Agree to use adequate contraception to avoid pregnancy.
* Provide signed informed consent.

Exclusion Criteria:

* Have any coagulation disorder other than hemophilia A or B.
* Treat with prophylactic treatment of coagulation factor.
* Treat with anticoagulant within 7d of the time of study drug administration.
* Have a history of arterial and/or venous thromboembolic events.
* Have platelet <100,000/mL,hemoglobin<90g/L.
* Severe liver or kidney disease.
* Bleeding in the central nervous system or throat before screening.
* Accept major operation or blood transfusion within 1 month of the time of screening.
* HIV positive with current CD4+ count of less than 200/μl.
* Have a known allergy to Blood product.
* Participate in other clinical research within 1 month of the time of study drug administration.
* Treat with coagulant within 7d of the time of study drug administration.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-29 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | From day 0 to up to day 8
Proportion of successfully treated bleeding episodes | 24 hours after administration of study drug

SECONDARY OUTCOMES:
Proportion of bleeding episodes with clinical relief of signs and symptoms | 4 hours、8 hours、24 hours after first administration of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, Ph.D, Principal Investigator — Hospital of Hematology, Chinese Academy of Medical Sciences
Locations (1):
- Hospital of Hematology, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu W, Zhou H, Huang R, Du X, Wang P, Zhou Z, Zheng C, Lou S, Ma J, Song Y, Dai X, Wang X, Yang R, Zhang L. A specific FX activator for bleeding treatment in hemophilia with inhibitors: multicenter, open-label, phase I/II trials. Blood Adv. 2026 Feb 4:bloodadvances.2025019486. doi: 10.1182/bloodadvances.2025019486. Online ahead of print. PMID 41637644
- [Derived] Liu W, Xue F, Fu R, Ding B, Li M, Sun T, Chen Y, Liu X, Ju M, Dai X, Wu Q, Zhou Z, Yu J, Wang X, Zhu Q, Zhou H, Yang R, Zhang L. Preclinical studies of a factor X activator and a phase 1 trial for hemophilia patients with inhibitors. J Thromb Haemost. 2023 Jun;21(6):1453-1465. doi: 10.1016/j.jtha.2023.01.040. Epub 2023 Feb 14. PMID 36796484